CLINICAL TRIAL: NCT01445587
Title: An Open-Label, Single Arm, Phase Ib/II Study of GSK2110183 in Subjects With Proteasome Inhibitor Refractory Multiple Myeloma
Brief Title: A Study of GSK2110183 in Subjects With Proteasome Inhibitor Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on the clinical activity, not safety data, of the AKT inhibitor, GSK has decided at this time to suspend further development of GSK2110183 as monotherapy.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115340
Record Dates: First submitted 2011-08-25; First posted 2011-10-04 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Cancer
Keywords: bortezomib; AKT inhibitor; multiple myeloma; GSK2110183; hematologic malignancies
MeSH Terms: conditions — Neoplasms; Multiple Myeloma; Hematologic Neoplasms | interventions — GSK2110183

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2110183 (Experimental): The oral dose of GSK2110183 the subjects received will be dependent on when the subject is enrolled to the study. GSK2110183 will be provided in 25mg and 50mg capsules containing the hydrochloride salt form of the API, microcrystalline cellulose, magnesium stearate, and microcrystalline cellulose (optional). They are filled into hard gelatin capsules. The 25mg tablets are opaque, swedish orange, size 2 capsules with no external markings, filled with a white powder. The 50mg tablets are opaque, white, size 1 capsules with no external markings, filled with a white powder.
  Interventions: Drug: Part 1; Cohort 1; Drug: Part 1; Cohort 2; Drug: Part 2; Stage 1; Drug: Part 2, Stage 2
- Bortezomib (Other): Bortezomib salvage therapy will be administered as a 3 to 5 second intravenous (IV) push at 1.3 mg/m2 on Days 1, 8, and 15 in each 21-day cycle until one of the Treatment Discontinuation Criteria is met.
  Interventions: Drug: Part 2; Stage 1; Drug: Part 2, Stage 2

INTERVENTIONS:
Drug: Part 1; Cohort 1 — On Cycle 0, Day -3, three subjects will be enrolled to receive a single oral dose of 125mg GSK2110183. After the 72 hour PK sampling is completed, the subjects will continue the 125mg GSK2110183 dose daily for 21 day cycles. If none of the 3 subjects experience one of the DLTs listed in the protocol during Cycle 1, the dose will be escalated to 150mg GSK2110183 for the subject enrolled to Cohort 2. Alternately, if 1 subject reports a DLT, then 3 more subjects will be enrolled at the same dose. If 2 of 6 subjects report a DLT, then the MTD has been exceeded. Subjects will remain on study until they meet one of the Treatment Discontinuation Criteria.
  Other Names: GSK2110183
  Arms: GSK2110183
Drug: Part 1; Cohort 2 — For Cohort 2, on Cycle 0, Day -3, three subjects will be enrolled to receive a single oral dose of 150mg GSK2110183. After the 72 hour PK sampling is completed, the subjects will continue the 150mg GSK2110183 dose daily for 21 day cycles. If none of the 3 subjects experience one of the DLTs listed in the protocol during Cycle 1, the MTD will be determined unless the PK and Pharmacodynamic data indicates another dose level should be evaluated. Alternately, if 1 subject reports a DLT, then 3 more subjects will be enrolled at the same dose. If 2 of 6 subjects report a DLT, then the MTD has been exceeded. Subjects will remain on study until they meet one of the Treatment Discontinuation Criteria.
  Other Names: GSK2110183
  Arms: GSK2110183
Drug: Part 2; Stage 1 — Following the completion of PK sampling and the determination of a Recommended Phase 2 Dose (RP2D) of GSK2110183 in Cohorts 1 and 2, subjects will be enrolled into Part 2, Stage 1 of the study. Twenty subjects will be enrolled in Stage 1. If no subject responds, the study will be stopped; otherwise, the study will continue enrollment of Stage 2.
  Other Names: GSK2110183+Bortezomib; GSK2110183
Drug: Part 2, Stage 2 — Twenty subjects will be enrolled in Part 2, Stage 2. If 4 or fewer of the 40 subjects (Stages 1 and 2) respond, the study will not be deemed as a success for GSK2110183 monotherapy. However, those subjects meeting the criteria for progression (as defined by IMWC Panel 1) who also meet the additional eligibility criteria for salvage therapy may proceed to GSK2110183 + bortezomib salvage therapy. GSK2110183 + bortezomib salvage therapy will be continued until one of the Treatment Discontinuation Criteria is met
  Other Names: GSK2110183; GSK2110183+Bortezomib

SUMMARY:
This is a single arm, open-label, Phase Ib/II study to evaluate the safety, pharmacokinetics, pharmacodynamics, and efficacy of the oral AKT inhibitor, GSK2110183, when administered to subjects with proteasome inhibitor refractory multiple myeloma (MM). During Part 1 of the study, GSK2110183 will be administered to subjects in sequential Pharmacokinetic (PK) Cohorts on a continuous daily dosing schedule in 21-day cycles until one of the Treatment Discontinuation Criteria is met. The PK Cohorts will characterize the PK of GSK2110183 in plasma and urine as well as determine the Recommended Phase 2 Dose (RP2D) of GSK2110183. The RP2D will be that dose that provides adequate PK exposure and biologic activity without exceeding the maximum tolerated dose (MTD) in MM subjects as defined in the current study. In Part 2 of the study, the RP2D will be further evaluated using a flexible 2-stage design with a stopping rule to allow for early termination based on lack of efficacy at the end of Stage 1. The first stage will accrue 20 subjects who will receive GSK2110183 at the RP2D. If a clinical response is observed in at least 1 subject in Stage 1, the study will proceed to Stage 2 and 20 additional subjects will be enrolled. GSK2110183 will be administered in Part 2 (Stage 1 and Stage 2) on a continuous daily dosing schedule in 21 day cycles until International Myeloma Working Group criteria for progression are met, at which point the subject will proceed to GSK 2110183 + bortezomib salvage therapy provided they meet the additional eligibility criteria for this phase of the study. GSK2110183 and bortezomib will be continued until one of the Treatment Discontinuation Criteria is met.

Exploratory PK/PD analyses may be performed to examine the potential relationships between GSK2110183 pharmacokinetics and pharmacodynamic biomarkers.

DETAILED DESCRIPTION:
This is a single arm, open-label, Phase Ib/II study to evaluate the safety, pharmacokinetics, pharmacodynamics, and efficacy of the oral AKT inhibitor GSK2110183 when administered to subjects with proteasome inhibitor refractory MM.

During Part 1 of the study, dose escalation will follow a 3 + 3 dose escalation procedure starting with an initial dosing regimen of 125 mg GSK2110183 with escalate to next dose level with an increase of GSK2110183 less than or equal to 50% if DLTs are below a certain level described in the protocol. Subjects will receive a single dose of GSK2110183 on Day -3 of Cycle 0, followed by PK sampling over the next 72 hours. Cycle 1 may commence at any time (but within 7 days) after collection of the 72 hour Cycle 0 PK sample. GSK2110183 will be administered to subjects in sequential PK Cohorts on a continuous daily dosing schedule in 21 day cycles until one of the Treatment Discontinuation Criteria is met. Sparse PK sampling will also be collected during the first 8 cycles. Urine PK samples will be collected prior to the first dose of GSK2110183 and as a 24-hour urine collection at steady-state. The PK Cohorts will characterize the pharmacokinetics of GSK2110183 in plasma and urine, as well as determine the RP2D of GSK2110183. The RP2D will be that dose that provides adequate PK exposure and biologic activity without exceeding the MTD in MM subjects as defined in the current study. GSK2110183 + bortezomib salvage therapy will not be given to subjects who progress on GSK2110183 monotherapy in the PK Cohorts. Following the completion of PK sampling in the PK Cohorts and the determination of a RP2D of GSK2110183, Part 2 of the study will then commence at the RP2D.

Part 2 of the study will further evaluate the R2PD using a flexible 2-stage design with a stopping rule to allow for early termination based on lack of efficacy at the end of Stage 1. GSK2110183 will be administered on a continuous daily dosing schedule in 21-day cycles until one of the Treatment Discontinuation Criteria is met. Twenty subjects will be enrolled in Stage 1, if no subject responds, the study will be stopped; otherwise, the study will continue to enroll an additional 20 subjects in Stage 2. At the end of Stage 2, if 4 or fewer of 40 subjects respond, the study will not be deemed as a success for the monotherapy. Those subjects meeting the criteria for progression during Part 2 [as defined by the 2011 Report of the International Myeloma Workshop Consensus Panel 1], who also meet the additional eligibility criteria for salvage therapy may proceed to GSK2110183 + bortezomib salvage therapy. GSK2110183 + bortezomib salvage therapy will be continued until one of the Treatment Discontinuation Criteria is met.

Exploratory PK/PD analyses may be performed in Part 1 and Part 2 to examine the potential relationships between GSK2110183 pharmacokinetics and pharmacodynamic biomarkers (e.g., pAKT, pPRAS40 in the bone marrow), markers for disease activity in serum (e.g., beta-2 microglobulin, C-reactive protein), or blood-based cytokines and angiogenesis factors (e.g., IL-6, VEGF).

A secondary objective of this study is to determine whether the addition of bortezomib to GSK2110183 has clinical activity in patients refractory to proteasome inhibitor therapy who progress on single-agent GSK2110183 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Male or female who is at least 18 years of age or older.
* Histologically confirmed diagnosis of secretory MM (must have measurable M protein in serum or urine) with one or more of the following:

Serum M-protein count greater than or equal to 1 g/dL Urinary M-protein greater than or equal to 200 mg/24 hours Serum free light chain (FLC) assay: involved FLC level greater than or equal to 10 mg/dL (greater than or equal to 100 mg/L) and a serum FLC ratio outside of normal range. Biopsy proven plasmacytoma

* Relapsed after 2 or more lines of systemic therapy including at least one proteasome inhibitor (i.e., bortezomib, carfilzomib) and at least one immunomodulatory agent (i.e., lenalidomide, pomalidomide) AND refractory to proteasome inhibitor therapy. Subjects will be considered refractory to proteasome inhibitor therapy if they experienced stable disease or progressive disease as the best response on their last proteasome inhibitor containing therapy OR progressed within 60 days following two or more cycles of proteasome inhibitor therapy. A line of therapy is generally separated by disease progression from a preceding line of therapy; therefore, the preparative regimen (with or without total body irradiation) and subsequent autologous stem cell rescue used for an autologous stem cell transplant are considered as one line of therapy.
* Subjects with a history of autologous stem cell transplant are eligible for study participation provided the following eligibility criteria are met:

Transplant was more than 100 days prior to study enrolment No active infection Subject meets the remainder of the eligibility criteria

* Performance status score of 0 to 2 according to Eastern Cooperative Oncology Group (ECOG).
* Able to swallow and retain oral medication.
* Fasting serum glucose less than126 mg/dL (<7 mmol/L). Subjects diagnosed previously with diabetes mellitus type 2 must also meet the additional following criteria:

Diagnosis of diabetes greater than 6 months prior to enrollment Glycosylated hemoglobin A1c (HbA1c) less than 8% at screening

* A female subject is eligible to participate if she is of the following:

Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) defined as premenopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone greater than 40 MlU/ml and estradiol less than 40 pg/ml (less than 147 pmol/L) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods listed in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

Childbearing potential, has a negative serum pregnancy test during the screening period, and agrees to use adequate contraception (methods listed in the protocol) from screening until four weeks after the last dose of GSK2110183. Note: Oral contraceptives are not reliable due to potential drug-drug interaction.

* Male subjects with female partners of childbearing potential must have had a prior vasectomy or agree to use adequate contraception from the time of the first dose of GSK2110183 until 3 months after the last dose of GSK2110183.
* Adequate organ function as defined by laboratory results within specific value ranges listed in the protocol.

Inclusion criteria: Salvage Therapy with GSK2110183 and Bortezomib:

* Platelet count greater than or equal to 70 X 10^9/L
* A subject whose ANC is greater than 1000/mm^3 before GSK2110183 monotherapy but whose ANC decreases below 1000/mm^3 at the time of transitioning to the salvage therapy is allowed up to 14 days following interruption of GSK2110183 dosing for ANC to recover to greater than or equal to 1000/mm^3.

Exclusion Criteria:

* Chemotherapy, radiotherapy, immunotherapy, or other anti-myeloma therapy within 14 days prior to the first dose of GSK2110183. In addition, any drug-related toxicity, except for alopecia, should have recovered to Grade 1 or less.
* Use of an investigational drug within 14 days or 5 half-lives, whichever is longer, preceding the first dose of GSK2110183.
* History of an allogeneic stem cell transplant. Subjects with a history of an autologous stem cell transplant are NOT excluded if they meet Inclusion Criterion 5 (Subjects with a history of autologous stem cell transplant are eligible for...).
* Current use of a prohibited medication.
* Current use of oral corticosteroids, with the exception of inhaled or topical corticosteroids.
* Anticoagulants (e.g., warfarin, low molecular weight heparin, direct thrombin inhibitors) at therapeutic doses or at low doses (e.g., prophylactic) are permitted only if the subject meets the partial thromboplastin time (PTT) and international normalization ratio (INR) entry criteria. Anticoagulant use must be monitored in accordance with local institutional practice.
* Presence of active GI disease or other condition that could affect GI absorption (e.g., malabsorption syndrome) or predispose subject to GI ulceration.
* Any major surgery within the last 14 days.
* Unresolved toxicity (except alopecia) greater than or equal to Grade 2 National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI-CTCAE v4) from previous anticancer therapy.
* Presence of greater than Grade 1 peripheral neuropathy.
* Type 1 diabetes mellitus.
* Any serious or unstable pre-existing medical, psychiatric, or other condition (including laboratory abnormalities) that could interfere with subject's safety or providing informed consent.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease, unstable hypertension).
* History of known human immunodeficiency virus infection.
* Subjects with a positive test for hepatitis B surface antigen or a positive test for hepatitis C antibody are excluded, regardless of the viral load. If hepatitis C antibody is positive, a confirmatory RIBA test may be performed. If the RIBA test is negative, the subject is eligible for the study.
* Primary or metastatic malignancy of the central nervous system.
* Diagnosis of or treatment for another malignancy within 2 years of enrollment, with the exception of complete resection of basal carcinoma or squamous cell carcinoma of the skin, or an in situ malignancy.
* QTC interval greater than or equal to 470 msec. NOTE: If initial result is prolonged, eligibility will be based on the average of manually calculated QTcF value from 3 ECGs (e.g., obtain 2 more ECGs at least 5 minutes apart and calculate the average of triplicate ECGs).
* Other clinically significant ECG abnormalities including 2nd degree (Type II) or 3rd degree atrioventricular block.
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within the past 6 months.
* Class III or IV heart failure as defined by the New York Heart Association [NYHA, 1994] functional classification system.
* Known hypersensitivity to GSK2110183, bortezomib, boron, and/or mannitol.
* Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of GSK2110183 in subjects with proteasome inhibitor refractory MM. | Subjects will continue on the study from the date of randomization until the date of the first documented progression or when the subjects meet one of the Treatment Discontinuation Criteria and may be assessed on average up to 48 months.
  Subjects with proteasome inhibitor refractory MM enrolled into Parts 1 and 2 will be evaluate for safety and tolerability of GSK2110183 by the assessment of adverse events and changes from baseline in safety assessments including laboratory parameters, vital signs, and electrocardiogram (ECG) parameters.
Determine a Recommended Phase II Dose (RP2D). | Subjects will continue on the study from the date of randomization until the date of the first documented progression or when the subjects meet one of the Treatment Discontinuation Criteria and may be assessed on average up to 48 months.
  RP2D is defined as a dose that provides adequate pharmacokinetics exposure and biologic activity without exceeding the Maximum Tolerated Dose (MTD) in Multiple Myeloma (MM) subjects as defined in the current study. RP2D will be defined in Part 1 of the study. The specific number of subjects to be enrolled is dependent on the number of Dose Limiting Toxicities (DLTs) reported; however, enrollment of approximately 18 subjects is estimated. The RP2D chosedn in Part 1 will be the dosing regimen used in Part 2.
Assess the clinical activity of GSK2110183 in subjects with proteasome inhibitor refractory MM. | Subjects will continue on the study from the date of randomization until the date of the first documented progression or when the subjects meet one of the Treatment Discontinuation Criteria and may be assessed on average up to 48 months.
  Subjects enrolled into Parts 1 and 2 will be assessed for overall response rate of GSK2110183 in subjects with proteasome inhibitor refractory Multiple Myeloma using the 2011 recommendations in the Report of the International Myeloma Workshop Consensus.

SECONDARY OUTCOMES:
Evaluate progression-free survival (PFS), overall survival (OS), time to response, and duration of response. | Subjects will continue on the study from the date of randomization until the date of the first documented progression or when the subjects meet one of the Treatment Discontinuation Criteria and may be assessed on average up to 48 months.
  Subjects enrolled into Parts 1 and 2 will be assessed for PFS, OS, time to response, and duration of response using the 2011 Report of the International Myeloma Workshop Consensus Panel 1. PFS is measured from the date of first dose until the date of disease progression or death due to any cause. OS is defined as the time from the date of first dose until the date of death due to any cause. Duration of response will be defined as the time from the first documented evidence of partial, very good partial, complete, or stringent complete tumor response until date of disease progression or death
Characterize the pharmacokinetics (PK) profile of GSK2110183 in subjects with proteasome inhibitor refractory MM. | Part 1: plasma PK on C0 (D-3), C1 (D15) pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 10-12, 14-22, 24, 48, and 72. In C2-8 (D1) pre-dose and post-dose. Urine PK on: C0 (D-3) pre-dose and C1 (D15) 24h post. Part 2: plasma PKs on C2-8 (D1) pre-dose and 1-2 hours post
  To characterize GSK2110183 pharmacokinetic parameters; area of concentration under the curve (AUC), Pre-dose (trough) concentration at the end of the dosing interval (Cτ), maximum observed concentration (Cmax), time of occurrence of Cmax (tmax) will be evaluated in the plasma and urine samples. The main PK sampling will take place in Part 1 of the study and Part 2 will have only sparse PK sampling.
Evaluate the clinical benefit of GSK2110183+bortezomib as salvage therapy for those subjects who progressed on GSK2110183 monotherapy. | Subjects will continue on the study from the date of randomization until the date of the first documented progression or when the subjects meet one of the Treatment Discontinuation Criteria and may be assessed on average up to 48 months.
  In Part 2 of the study, subjects whom bortezomib is added to GSK2110183 due to disease progression on GSK2110183 monotherapy overall response rate (ORR = stringent complete response + complete response + very good partial response + partial response rates), PFS, duration of response, and time-to-next-therapy will be evaluated.
Explore the association of biologic/clinical endpoints with DNA or protein profiles from malignant cells as data permit. | Assessed up to 48 months.
  Subjects enrolled into Parts 1 and 2 will have samples collected for analysis of the markers of AKT pathway activation (e.g., pAKT, pPRAS40) in bone marrow biopsy and/or aspirate samples, potential predictive markers of response (e.g., cytogenetics, FISH, Ki67, mutations in NRAS and KRAS) in bone marrow biopsy and/or aspirate samples, and soluble cytokine levels (e.g., VEGF, IL-6, IGF1) in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Melbourne, Victoria, Australia